CLINICAL TRIAL: NCT02586896
Title: Comparing Interventions for Opioid Dependent Patients Presenting in Medical Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-00862
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Mass Screening; Restraint, Physical; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengths-based Case Management (SBCM) (Experimental): The structure of SBCM follows the widely accepted functions of case management-assessment, planning, linking, monitoring and advocacy-and the theory-driven gestalt of the strengths perspective. Strengths-based principles include an emphasis on client strengths, teaching clients a method for setting and completing goals, and development of a strong working alliance.
  Interventions: Behavioral: Strengths-based Case Management (SBCM)
- Screening, Assessment and Referral (SAR) (Active Comparator): Following randomization, participants in the SAR condition will be provided with minimal scripted feedback to let them know that their assessment indicates substance dependence, and given a recommendation to seek treatment.
  Interventions: Behavioral: Screening, Assessment, and Referral (SAR)

INTERVENTIONS:
Behavioral: Strengths-based Case Management (SBCM) — The six case management sessions for the proposed trial are based on those described in manuals developed by Dr. Rapp for two clinical trials, one supported by National Institute on Drug Abuse (NIDA) and another by the Centers for Disease Control (CDC). Each session is guided by specific objectives that promote linkage with and retention in substance abuse treatment, particularly pharmacotherapy for opioid dependence in a specialty or primary care setting. Objectives from the earlier trials will be adapted to fit the specific context of this trial, linking with and staying in treatment following an emergency department visit. Initiation of the relationship between client and case manager begins immediately following random assignment and termination takes place when either (1) six sessions have occurred; (2) ninety days have elapsed; or (3) clients discontinue involvement.
  Arms: Strengths-based Case Management (SBCM)
Behavioral: Screening, Assessment, and Referral (SAR) — The research assistant will provide these participants with an information sheet listing treatment (including both specialty treatment centers and primary care clinics that provide buprenorphine) and self-help resources in their community. The referral sheet includes names, addresses, and phone numbers of local addiction treatment agencies. Because the emergency department does not currently screen or refer systematically, the SAR condition represents a level of care significantly higher than "treatment as usual." Participants will also receive an informational pamphlet about drug use and its consequences, addiction, and treatment.
  Arms: Screening, Assessment and Referral (SAR)

SUMMARY:
This study will compare the effects of brief strengths-based case management (SBCM) to the effects of screening, assessment and referral alone (SAR) in opioid-dependent patients. Participants meeting DSM-IV criteria for opioid dependence will be randomly assigned (150 per group) to receive 1) up to 6 sessions of SBCM; or 2) SAR. Follow-up assessments will be completed at 3 and 6 months, by staff who are blinded to treatment condition.

DETAILED DESCRIPTION:
As addiction treatment becomes increasingly integrated into the medical care system, two models have rightly received a great deal of attention. The first is the use of Screening, Brief Intervention, and Referral to Treatment (SBIRT) models to identify cases, provide therapeutic contact, and refer the more severe cases to longer-term care. The second is the treatment of addictions using medical models of treatment, including those that can be implemented in primary care settings. Much less attention has been paid to optimizing strategies for bridging the gap between SBIRT and more intensive/longer-term treatment for those on the severe end of the spectrum. This factor is of critical importance for opioid dependent patients, whose needs are not met by brief interventions or brief treatment. Emergency room interventions for substance use disorders have been largely limited to brief interventions/SBIRT models, and these have focused primarily on alcohol. Although there is a substantial literature documenting the value of case management in linking drug users to treatment, this approach has not been applied to drug users in the emergency department (ED) setting.

In a sample of opioid dependent patients seen in a medical ED who are not currently engaged in treatment, this study will compare the effects of brief strengths-based case management (SBCM) to the effects of screening, assessment and referral alone. Participants meeting DSM-IV criteria for opioid dependence will be randomly assigned (150 per group) to receive 1) Screening, Assessment and Referral or 2) up to 6 sessions of SBCM based on the model previously implemented by Rapp and colleagues in prior studies. Staff who are blinded to treatment condition will complete follow-up assessments at 3 and 6 months. Aims of the study are to identify the main effects of SBCM on substance abuse treatment initiation and engagement, use of opioids and other drugs, and broader measures of health and life functioning; to examine the interactions between treatment assignment and selected participant attributes in predicting treatment initiation, engagement, and substance use outcomes; and to examine effects of treatment involvement on substance use outcomes in the two treatment groups.

The proposed study will be the first trial using a case management approach to link drug dependent patients presenting in EDs to longer-term addiction treatment. It will be one of the first trials focusing specifically on opioid dependent patients in medical EDs. A further innovative feature is that the case management approach will emphasize linkage to pharmacotherapy, facilitating linkage to office-based buprenorphine, methadone, or naltrexone for patients who desire this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Registration as patient in the ED during study screening hours;
2. Endorsement of three or more opioid dependence criteria on the DSM-IV checklist
3. Age 18 years or older;
4. Adequate English proficiency;
5. Ability to provide informed consent;
6. Self-report use of opioids in the last 30 days

Exclusion Criteria:

1. Inability to participate due to emergency treatment;
2. Significant impairment of cognition or judgment rendering the person incapable of informed consent. (e.g., traumatic brain injury, delirium, intoxication);
3. Status as a prisoner or in police custody at the time of treatment;
4. Current engagement in substance use disorder treatment;
5. Residence more than 50 miles from the location of follow-up visits;
6. Inability to provide sufficient contact information (must provide at least 2 reliable locators);
7. Unavailable for follow-up (e.g., planning to relocate within 6 months)
8. Prior participation in the current study.
9. Current participation in a research study related to substance use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Bogenschutz, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- Bellevue Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Regis A, Meyers-Ohki SE, Mennenga SE, Greco PP, Glisker R, Kolaric R, McCormack RP, Rapp RC, Bogenschutz MP. Implementation of strength-based case management for opioid-dependent patients presenting in medical emergency departments: rationale and study design of a randomized trial. Trials. 2020 Sep 3;21(1):761. doi: 10.1186/s13063-020-04684-6. PMID 32883337

RESULTS

PARTICIPANT FLOW:
Groups:
- Strengths-based Case Management (SBCM): The structure of SBCM follows the widely accepted functions of case management-assessment, planning, linking, monitoring and advocacy-and the theory-driven gestalt of the strengths perspective. Strengths-based principles include an emphasis on client strengths, teaching clients a method for setting and completing goals, and development of a strong working alliance.
  The six case management sessions for this trial were based on those described in manuals developed by Dr. Rapp for two previous clinical trials. Each session was guided by specific objectives that promote linkage with and retention in substance abuse treatment, particularly pharmacotherapy for opioid dependence. Initiation of the relationship between client and case manager began immediately following random assignment and termination took place when either (1) six sessions had occurred; (2) ninety days had elapsed; or (3) clients discontinued involvement.
- Screening, Assessment and Referral (SAR): Participants in the SAR condition were provided with minimal scripted feedback to let them know that their assessment indicates substance dependence, and given a recommendation to seek treatment. The research assistant provided SAR participants with an information sheet listing treatment (including both specialty treatment centers and primary care clinics that provide buprenorphine) and self-help resources in their community. The referral sheet included names, addresses, and phone numbers of local addiction treatment agencies. Participants also received an informational pamphlet about drug use and its consequences, addiction, and treatment.
  Because the emergency department does not currently screen or refer systematically, the SAR condition represented a level of care significantly higher than "treatment as usual."
Period: Overall Study
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
Started | 150 | 150
3-Month Follow-up | 126 | 123
Completed (6-Month Follow-Up) | 131 | 133
Not Completed | 19 | 17

BASELINE CHARACTERISTICS:
Population: 2 SBCM participants excluded from analysis (1 determined ineligible; 1 pilot SBCM participant); 1 SAR participant excluded from analysis (withdrawn)
Groups:
- Strengths-based Case Management (SBCM): Participants received up to six sessions of Strengths-based Case Management (SBCM) within 90 days of randomization.
- Screening, Assessment and Referral (SAR): Participants received a detailed referral sheet, an informational pamphlet, and scripted feedback recommending they seek treatment.
- Total: Total of all reporting groups
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR) | Total
Number analyzed (Participants) | 148 | 149 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (10.8) | 43.0 (10.8) | 43.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 130 | 126 | 256
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1 | 1 | 2
  Asian, Asian-American/Pacific Islander | 3 | 5 | 8
  Black or African American | 47 | 50 | 97
  Hispanic, Cuban | 1 | 0 | 1
  Hispanic, Mexican | 0 | 0 | 0
  Hispanic, New Mexican/Spanish-American | 0 | 4 | 4
  Hispanic, Puerto Rican | 43 | 33 | 76
  Hispanic, Other Latin American | 8 | 9 | 17
  White, not of Hispanic origin | 36 | 38 | 74
  Other ethnic group | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Initiation of Treatment for Opioid Dependence
Description: "Initiation" is defined as a dichotomous outcome (yes/no), and is considered to have occurred if patients report any substance abuse counseling sessions (excluding SBCM) from the time of the baseline assessment up to the day before the three-month interview, as captured via self-report on the Form 90-D.
Time Frame: 3 months
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Groups:
- Strengths-based Case Management (SBCM): Strengths-based Case Management (SBCM)
- Screening, Assessment and Referral (SAR): Screening, Assessment and Referral (SAR)
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
Number analyzed (Participants) | 148 | 149
Participants
  Initiated | 85 | 74
  Did Not Initiate | 63 | 75

2. Primary Outcome: Engagement in Treatment for Opioid Dependence
Description: Using the same timeframe as "initiation," "engagement" is defined as the number days of medication use for opioid dependence, based on Form 90-D self-report verified by clinic dosing logs and Prescription Drug Monitoring Program records.
Time Frame: 3 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: % days
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
Number analyzed (Participants) | 148 | 149
% days | 21.77 (35.07) | 17.72 (30.99)
Statistical Analysis 1: Comparison: Strengths-based Case Management (SBCM) vs Screening, Assessment and Referral (SAR); Test type: Superiority; p = 0.29, ANOVA

3. Secondary Outcome: Number of Participants With Successful Outcome for Opioid Use
Description: "Successful outcome" will be defined as 1) 3-month urine negative for opioids (opiates, oxycodone, methadone, buprenorphine, or propoxyphene) unless prescribed for opioid dependence, and 2) no more than two days of self-reported opioid use on the Form 90-D in the 4 weeks (30 days) prior to the 3-month evaluation.
Time Frame: 3 months
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
Number analyzed (Participants) | 148 | 149
Participants
  Successful outcome | 41 | 28
  No successful outcome | 107 | 121

4. Secondary Outcome: Score on World Health Organization Quality of Life (WHOQoL) Brief Questionnaire
Description: The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. Participants express how much they have experienced the items in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). Raw domain score is the sum of respective item scores. All domain scores are reported between 4 and 20.
Time Frame: 3 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
Number analyzed (Participants) | 148 | 149
units on a scale | 11.23 (4.61) | 11.22 (4.45)
Statistical Analysis 1: Comparison: Strengths-based Case Management (SBCM) vs Screening, Assessment and Referral (SAR); Test type: Superiority; p = 0.91, ANOVA

5. Secondary Outcome: Initiation in Participants With Higher Levels of Environmental Instability at Baseline
Description: as for outcome 1
Time Frame: 3 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: % of participants
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
Number analyzed (Participants) | 148 | 149
% of participants | 62.5 (7.8) | 57.8 (7.2)
Statistical Analysis 1: Comparison: Strengths-based Case Management (SBCM) vs Screening, Assessment and Referral (SAR); Test type: Superiority; p = 0.09, ANOVA

6. Secondary Outcome: Engagement in Participants With Higher Levels of Environmental Instability at Baseline
Description: as for outcome 2
Time Frame: 3 months
Measure: Mean (Standard Error); unit: % days
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
Number analyzed (Participants) | 148 | 149
% days | 22.16 (5.21) | 19.89 (4.76)
Statistical Analysis 1: Comparison: Strengths-based Case Management (SBCM) vs Screening, Assessment and Referral (SAR); Test type: Superiority; p = 0.54, ANOVA

ADVERSE EVENTS:
Time Frame: Consent through final 6-month follow-up
Description: Events not meeting the study definition of AE:
  * Mild unrelated event
  * Moderate unrelated event
  * Substance use events (e.g., worsening drug use, need for higher level of care, withdrawal symptoms, craving, related medical events)
  Events not meeting the study definition of SAE:
  * Admission for drug detox/treatment
  * Admission for preplanned surgeries
  * Admission for scheduled labor/delivery
  * Admission for a medical event, unless severe, life threatening, or resulting in death
Arm/Group | Strengths-based Case Management (SBCM) | Screening, Assessment and Referral (SAR)
All-Cause Mortality (participants affected / at risk) | 4/150 | 1/150
Serious Adverse Events (participants affected / at risk) | 17/150 | 8/150
Other Adverse Events (participants affected / at risk) | 3/150 | 2/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strengths-based Case Management (SBCM) (N=150) | Screening, Assessment and Referral (SAR) (N=150)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Death (cause unknown) (General disorders) | 3 (3) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 10 (11) | 5 (6)
Withdrawal of life support (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strengths-based Case Management (SBCM) (N=150) | Screening, Assessment and Referral (SAR) (N=150)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT02586896/Prot_SAP_000.pdf